CLINICAL TRIAL: NCT01007032
Title: A Phase 1 Study Evaluating the Safety and Pharmacokinetic Profiles of IMC-A12 Administered Every 2 Weeks or Every 3 Weeks to Japanese Patients With Advanced Solid Tumors
Brief Title: A Study of IMC-A12 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Parexel (Industry); Medidata Solutions (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 13905; 21-1258 (Other: PMDA (MoH) in Japan); CP13-0813 (Other: ImClone Systems); I5A-IE-JAEA (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-10

CONDITIONS: Tumors
Keywords: anti-IGF-IR; monoclonal; solid tumor; insulin-like growth factor
MeSH Terms: conditions — Neoplasms | interventions — cixutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cixutumumab (Experimental): Participants receive IV cixutumumab every 2 or 3 weeks. A cycle equals 6 weeks, with radiological evaluation of tumor response after each cycle. After 1st cycle, pts with a complete response (CR), PR, or SD continue to receive cixutumumab cohort dose and schedule disease progression. 3 pts enroll in each cohort. Starting dose in Cohort 1 is 6 mg/kg every 2 weeks. Dose escalation from Cohort 1 to Cohort 2 (10 mg/kg every 2 weeks) occurs at least 3 pts in Cohort 1 completes 1 cycle of therapy. Enrollment into Cohort 3 (starting dose: 15 mg/kg administered every 3 weeks) will not proceed until at least 3 pts have completed one cycle of therapy in Cohort 2. Pts enroll in Cohort 4 once at least 3 pts have completed once cycle of therapy in Cohort 3; pts in Cohort 4 receive 20 mg/kg every 3 weeks.
  Interventions: Biological: Cixutumumab

INTERVENTIONS:
Biological: Cixutumumab — Cixutumumab intravenously
  Other Names: IMC-A12; LY3012217

SUMMARY:
In this study, participants will initially receive intravenous (IV) cixutumumab (IMC-A12) every 2 weeks or every 3 weeks for 6 weeks (one cycle). After the first cycle, participants experiencing a best overall response of complete response, partial response, or stable disease will continue to receive cixutumumab at their cohort dose and schedule until there is evidence of progressive disease (PD), or until other withdrawal criteria are met. Participants will be enrolled at one study center, located in the National Cancer Center Hospital - East, Kashiwa, Japan. Approximately 20-30 participants are anticipated.

DETAILED DESCRIPTION:
Participants in this single-center, open-label, dose-escalation, Phase 1 study will initially receive intravenous (IV) cixutumumab every 2 weeks or every 3 weeks for 6 weeks (one cycle). After the first cycle, participants experiencing a best overall response of complete response (CR), partial response (PR), or stable disease (SD) will continue to receive cixutumumab at their cohort dose and schedule until there is evidence of progressive disease (PD), or until other withdrawal criteria are met.

A minimum of three participants will be enrolled in each cohort. The starting dose in Cohort 1 will be 6 mg/kg, administered every 2 weeks. Dose escalation from Cohort 1 to Cohort 2 (10 mg/kg administered every 2 weeks) will occur once at least three participants in Cohort 1 have completed one cycle of therapy (ie, completed the initial 6 week treatment period or discontinued therapy due to an cixutumumab - related adverse event [AE]).

Enrollment into Cohort 3 (starting dose: 15 mg/kg administered every 3 weeks) will not proceed until all participants have completed one cycle of therapy (as defined above) in Cohort 2. Similarly, participants will be enrolled in Cohort 4 once at least three participants have completed one cycle of therapy in Cohort 3;participants in Cohort 4 will receive 20 mg/kg administered every 3 weeks. Toxicity data for each cohort will be reviewed prior to any dose escalation. No intrapatient dose escalation is permitted. Participants in any cohort who do not complete the first 6 weeks of treatment for reasons other than an cixutumumab-related toxicity will be replaced.

A dose-limiting toxicity (DLT) is defined as one of the following events, if considered by the investigator to be definitely, probably, or possibly related to cixutumumab: Grade 4 neutropenia lasting > 7 days; Grade 4 anemia; Grade ≥ 3 thrombocytopenia; Grade ≥ 3 neutropenia associated with fever; Grade 3 or 4 nonhematologic toxicity, excluding electrolyte abnormality and Grade 3 hyperglycemia; Grade 4 hyperglycemia; and/or Grade 4 or uncontrollable hypertension.

If three participants complete the first 6-week cycle (according to the definition outlined above) with no DLTs, dose escalation to Cohort 2 may proceed. If one DLT is observed in the initial three participants of Cohort 1 (or any cohort) during Cycle 1, three additional participants will be enrolled into that cohort. If no additional DLTs are observed, dose escalation may continue as described above.

If two or more participants in Cohort 1 experience a DLT, six participants will be enrolled into Cohort 1A (receiving 4 mg/kg every 2 weeks). If two or more participants experience a DLT in dose Cohort 3, six participants will be enrolled into dose Cohort 3A (10 mg/kg every 3 weeks). If two or more participants experience a DLT in dose Cohorts 2 or 4, six additional participants will be enrolled into the previous cohort (Cohort 1 or Cohort 3, respectively), and the previous cohort will be considered the maximum tolerated dose for that dosing schedule. If two or more participants in any cohort experience a DLT on Week 7 or beyond (after Cycle 1), the data will be reviewed and enrollment may be suspended. The Sponsor and Principal Investigator, with reference to the review of the Independent Data Safety Evaluation Committee (established in a separate document), will determine whether enrollment should resume.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor participant who has been histopathologically or cytologically documented
* Advanced primary or recurrent solid tumor participant who has not responded to standard therapy or for whom no standard therapy is available
* The participant has measurable or nonmeasurable lesions according to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.0) guidelines
* The participant has an Eastern Cooperative Oncology Group performance status (ECOG PS)score of 0-1 at study entry
* The participant is able to provide informed consent
* The participant is age 20 years or older
* The participant has a life expectancy of > 3 months
* The participant has adequate hematologic function, as defined by:
* An absolute neutrophil count (ANC) ≥ 1500/m3 or /μL
* A hemoglobin ≥ 10 g/dL; and
* A platelet count ≥ 100,000/mm3 or /μL
* The participant has adequate hepatic function, as defined by:
* Total bilirubin ≤ 1.8 mg/dL
* Aspartate transaminase (AST) ≤ 2.5 times the upper limit of site-specific normal ranges (five times in case of liver metastasis)
* Alanine transaminase (ALT) ≤ 2.5 times the upper limit of site-specific normal ranges (five times in case of liver metastasis)
* The participant has adequate renal function, as defined by:
* Serum creatinine ≤ 1.5 mg/dL
* Calculated serum creatinine clearance (Cockcroft-Gault) ≥ 60 mL/min
* The participant has fasting blood sugar < 120 mg/dL or below the institutional upper limit of normal (ULN) before study entry (one retest of an elevated level is permitted at the discretion of the investigator)
* The participant has adequate coagulation function, as defined by an international normalized ratio (INR) ¬ 1.5
* The participant agrees to use adequate contraception for the duration of study participation and for 12 weeks after the last dose of study therapy.
* The participant has adequate recovery from recent surgery, chemotherapy, and radiation therapy (including palliative radiation therapy). At least 28 days (6 weeks for nitrosoureas or mitomycin C) must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent or device, or prior radiation therapy. For treatment with unapproved monoclonal antibodies, a minimum of 8 weeks must have elapsed
* The participant is willing to comply with study procedures until the end of therapy

Exclusion Criteria:

* The participant has received chemotherapy or therapeutic radiotherapy within 28 days (6 weeks for nitrosoureas or mitomycin C) prior to entering the study, or the participant has ongoing side effects ≥ Grade 2 due to agents administered more than 28 days earlier
* The participant has undergone major surgery (eg,laparotomy, thoracotomy,removal of organ(s)) within 28 days prior to study entry, or subcutaneous venous access device placement within 7 days prior to study entry
* The participant has elective or planned surgery to be conducted during the trial
* The participant has documented and/or symptomatic brain or leptomeningeal metastases (participants who are clinically stable (no symptoms during the 4 weeks prior to enrollment) with an assessment that no further treatment (radiation, surgical excision, or administration of steroids) is required are permitted to enter the study)
* The participant has an uncontrolled intercurrent illness including, but not limited to:
* Thrombotic or hemorrhagic disorders
* Gross hemoptysis (approximately one-half a teaspoon)
* Ongoing or active infection requiring systemic antibiotic treatment
* Congestive heart failure (Class III or IV per the New York Heart Association classification for heart disease)
* Angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
* Uncontrolled hypertension (systolic blood pressure > 150 mm Hg, diastolic blood pressure > 95 mm Hg)
* Cardiac arrhythmia requiring treatment (NCICTCAE Version 3.0 Grade 3), or asymptomatic sustained ventricular tachycardia
* Peripheral neuropathy of any etiology ≥ Grade 2 (NCI-CTCAE Version 3.0); or
* Any other serious uncontrolled medical disorder(s) in the opinion of the investigator
* The participant has a serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to study entry
* The participant has experienced any Grade 3/4 gastrointestinal bleeding within 3 months prior to study entry
* The participant has participated in clinical studies of unapproved experimental agents or procedures within 4 weeks prior to study entry for small molecules, or 8 weeks prior to study entry for unapproved monoclonal antibodies
* The participant has received any previous treatment with agents targeting the insulin-like growth factor hormone (IGF-IR), approved or unapproved
* The participant has a known allergy to any of the treatment components (monoclonal antibodies or other therapeutic proteins such as fresh frozen plasma, human serum albumin, cytokines, or interleukins). In the event that there is suspicion the participant may have allergies, the participant should be excluded
* The participant, if female, is pregnant (confirmed by urine or serum pregnancy test) or lactating
* The participant has a known alcohol or drug dependency
* The participant is Hepatitis B Virus (HBV) antigen-, Hepatitis C Virus (HCV) antibody-, or HIV antibody-positive (asymptomatic healthy carriers with detectable HBV-DNA, HCV-RNA may be enrolled into the trial)
* The participant is assessed as inadequate for the study by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- ImClone Investigational Site, Kashiwa, Japan

REFERENCES:
- [Derived] Doi T, Shitara K, Kojima T, Yoshino T, Dontabhaktuni A, Rebscher H, Tang S, Cosaert J, Ohtsu A. A phase I study evaluating cixutumumab, a type 1 insulin-like growth factor receptor inhibitor, given every 2 or 3 weeks in Japanese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2016 Jun;77(6):1253-62. doi: 10.1007/s00280-016-3041-7. Epub 2016 Apr 30. PMID 27139036

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had progressive disease (PD) were considered to complete the study.
Groups:
- Cixutumumab Cohort 1: 6 milligrams/kilograms (mg/kg) of cixutumumab was administered intravenously (IV) every 2 weeks for 6 weeks (one cycle).
- Cixutumumab Cohort 2: 10 mg/kg of cixutumumab was administered IV every 2 weeks for 6 weeks (one cycle).
- Cixutumumab Cohort 3: 15 mg/kg of cixutumumab was administered IV every 3 weeks for 6 weeks (one cycle).
- Cixutumumab Cohort 4: 20 mg/kg of cixutumumab was administered IV every 3 weeks for 6 weeks (one cycle).
Period: Overall Study
Arm/Group | Cixutumumab Cohort 1 | Cixutumumab Cohort 2 | Cixutumumab Cohort 3 | Cixutumumab Cohort 4
Started | 4 | 7 | 3 | 7
Received at Least 1 Dose of Study Drug | 4 | 7 | 3 | 7
Completed | 4 | 6 | 2 | 6
Not Completed | 0 | 1 | 1 | 1
Not completed — On Study Treatment at Cut-off Date | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cixutumumab Cohort 1: 6 mg/kg of cixutumumab was administered IV every 2 weeks for 6 weeks (one cycle).
- Total: Total of all reporting groups
Arm/Group | Cixutumumab Cohort 1 | Cixutumumab Cohort 2 | Cixutumumab Cohort 3 | Cixutumumab Cohort 4 | Total
Number analyzed (Participants) | 4 | 7 | 3 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.52) | 60.5 (6.82) | 62.2 (5.57) | 60.3 (8.67) | 60.9 (7.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 2 | 3 | 9
  Male | 4 | 3 | 1 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 7 | 3 | 7 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 7 | 3 | 7 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 4 | 7 | 3 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Summary Listing of Percentage of Participants Reporting Treatment-Emergent Adverse Events
Description: A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: Up To 63 Months
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Cixutumumab Cohort 1: 6 mg/kg of cixutumumab was administered intravenously (IV) every 2 weeks for 6 weeks (one cycle).
Arm/Group | Cixutumumab Cohort 1 | Cixutumumab Cohort 2 | Cixutumumab Cohort 3 | Cixutumumab Cohort 4
Number analyzed (Participants) | 4 | 7 | 3 | 7
percentage of participants | 100 | 85.7 | 100 | 85.7

2. Primary Outcome: Number of Participants With a Dose Limiting Toxicity (DLT)
Description: DLTs were defined as any cixutumumab-related Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE 3.0) Grade 3 or 4 adverse events (reported in the subsequent Primary Outcome Measure).
Time Frame: First Dose Up to 6 Weeks
Population: All participants who completed the first cycle of 6 weeks or discontinued due to Dose Limiting Toxicities (DLTs).
Measure: Number; unit: participants
Groups:
- Cixutumumab 6 mg/kg: 6 mg/kg of cixutumumab was administered intravenously (IV) every 2 weeks for 6 weeks (one cycle).
- Cixutumumab 10 mg/kg: 10 mg/kg of cixutumumab was administered IV every 2 weeks for 6 weeks (one cycle).
- Cixutumumab 15 mg/kg: 15 mg/kg of cixutumumab was administered IV every 3 weeks for 6 weeks (one cycle).
- Cixutumumab 20 mg/kg: 20 mg/kg of cixutumumab was administered IV every 3 weeks for 6 weeks (one cycle).
Arm/Group | Cixutumumab 6 mg/kg | Cixutumumab 10 mg/kg | Cixutumumab 15 mg/kg | Cixutumumab 20 mg/kg
Number analyzed (Participants) | 4 | 7 | 3 | 7
participants | 0 | 0 | 0 | 0

3. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax)
Time Frame: Prior to Infusion and Immediately Following End of Infusion (Cohorts 1 and 2) at 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264 and 336 hours and (Cohorts 3 and 4) at 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264, 336, 408 and 504 Hours Following End of Infusion
Population: All participants who received at least 1 dose of study drug and had evaluable PK data for Cmax (First Dose and Fourth doses for Cohorts 1 and 2 and First and Third doses for Cohorts 3 and 4.)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Arm/Group | Cixutumumab Cohort 1 | Cixutumumab Cohort 2 | Cixutumumab Cohort 3 | Cixutumumab Cohort 4
Number analyzed (Participants) | 3 | 5 | 3 | 7
microgram/milliliter (μg/mL)
  First Dose | 184 (34) | 643 (95) | 1020 (32) | 1390 (22)
  Fourth Dose or Third Dose: number analyzed (Participants) | 1 | 3 | 0 | 1
  Fourth Dose or Third Dose | NA (NA) — The geometric mean and % coefficient of variation (CV) were not calculated because there was 1 evaluable participant. Cmax=390.019 μg/mL | 734 (102) |  | NA (NA) — The geometric mean and % CV were not calculated because there was 1 participant in Cohort 4. Cmax=1741.312 μg/mL

4. Primary Outcome: PK: Area Under the Curve From Zero to Infinity AUC(0-∞)
Time Frame: as for outcome 3
Population: All participants who received at least 1 dose of study drug and had evaluable PK data for AUC(0-∞). First Dose for Cohorts 1, 2, 3, and 4.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms•hour/milliliter (μg•h/mL)
Arm/Group | Cixutumumab Cohort 1 | Cixutumumab Cohort 2 | Cixutumumab Cohort 3 | Cixutumumab Cohort 4
Number analyzed (Participants) | 4 | 4 | 2 | 7
micrograms•hour/milliliter (μg•h/mL) | 26500 (19) | 42000 (50) | 120000 (51) | 157000 (26)

5. Secondary Outcome: Number of Participants With Serum Anti-Cixutumumab Antibody Assessment Immunogenicity
Description: No participants were analyzed for the development of circulating positive anti-cixutumumab antibodies due to no assay available.
Time Frame: 6 months
Population: No participants were analyzed due to no assay available.
Arm/Group | Cixutumumab Cohort 1 | Cixutumumab Cohort 2 | Cixutumumab Cohort 3 | Cixutumumab Cohort 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Primary Outcome: PK: Area Under Concentration Versus Time Curve During One Dosing Interval (AUCtau)
Time Frame: as for outcome 3
Population: All participants who received 1 dose of study drug and had evaluable PK data for (AUCtau). Fourth doses for Cohorts 1 and 2. No participant was evaluable in Cohorts 3 and 4.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (μg•h/mL)
Arm/Group | Cixutumumab Cohort 1 | Cixutumumab Cohort 2 | Cixutumumab Cohort 3 | Cixutumumab Cohort 4
Number analyzed (Participants) | 2 | 3 | 0 | 0
(μg•h/mL) | 36400 (8) | 63600 (40) |  |

7. Primary Outcome: Half-life (t1/2)
Time Frame: Prior to Infusion and Immediately Following End of Infusion (Cohorts 1 and 2) at 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264, and 336 hours and (Cohorts 3 and 4) at 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264, 336, 408 and 504 hours) Following End of Infusion
Population: All participants who received at least 1 dose of study drug and had evaluable PK data for t1/2 estimation (First Dose and Fourth doses for Cohorts 1 and 2 and First Dose and Third doses for Cohorts 3 and 4.)
Measure: Geometric Mean (Full Range); unit: day
Arm/Group | Cixutumumab Cohort 1 | Cixutumumab Cohort 2 | Cixutumumab Cohort 3 | Cixutumumab Cohort 4
Number analyzed (Participants) | 4 | 7 | 3 | 7
day
  First Dose: number analyzed (Participants) | 4 | 4 | 3 | 7
  First Dose | 6.08 [5.29 to 6.88] | 4.06 [3.33 to 6.04] | 9.88 [6.58 to 16.0] | 8.83 [4.67 to 13.8]
  Fourth Dose or Third Dose (n=2,2,1,0): number analyzed (Participants) | 2 | 2 | 1 | 0
  Fourth Dose or Third Dose (n=2,2,1,0) | NA [NA to NA] — The geometric mean and range were not calculated because there were 2 participants in Cohort 1. t1/2 values = 5.50; 4.75 days. | NA [NA to NA] — The geometric mean and range were not calculated because there were 2 participants in Cohort 2. t1/2 values = 4.29; 5.92 days. | NA [NA to NA] — The geometric mean and full range was not calculated due to 1 evaluable participant in Cohort 3. t1/2 value=6.96 days |

8. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR])
Description: Response defined per Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria: Complete Response (CR)=disappearance of all target lesions; Partial Response (PR)=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions.
Time Frame: From the First Dose up to 32 Months
Population: All participants who received 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cixutumumab Cohort 1 | Cixutumumab Cohort 2 | Cixutumumab Cohort 3 | Cixutumumab Cohort 4
Number analyzed (Participants) | 4 | 7 | 3 | 7
percentage of participants | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 16.1]

9. Primary Outcome: Drug Clearance (CL)
Time Frame: as for outcome 7
Population: All participants who received at least 1 dose of study drug and had evaluable PK data for CL estimation (First Dose and Fourth doses for Cohorts 1 and 2 and First Dose and Third doses for Cohorts 3 and 4.)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/h)
Arm/Group | Cixutumumab Cohort 1 | Cixutumumab Cohort 2 | Cixutumumab Cohort 3 | Cixutumumab Cohort 4
Number analyzed (Participants) | 4 | 7 | 3 | 7
Liter/hour (L/h)
  First Dose: number analyzed (Participants) | 4 | 4 | 2 | 7
  First Dose | 0.0137 (13) | 0.0135 (53) | NA (NA) — The geometric mean and CV were not calculated due to 2 participants in Cohort 3. Values=0.00574; 0.00948 L/h | 0.00709 (41)
  Fourth Dose or Third Dose (n=2,3,0,0): number analyzed (Participants) | 2 | 3 | 0 | 0
  Fourth Dose or Third Dose (n=2,3,0,0) | NA (NA) — The geometric mean and CV were not calculated due to 2 participants in Cohort 1. Values=0.0124; 0.0118 L/h | 0.00994 (49) |  |

ADVERSE EVENTS:
Description: All participants who received at least 1 dose of study drug.
Arm/Group | Cixutumumab Cohort 1 | Cixutumumab Cohort 2 | Cixutumumab Cohort 3 | Cixutumumab Cohort 4
Serious Adverse Events (participants affected / at risk) | 1/4 | 5/7 | 1/3 | 0/7
Other Adverse Events (participants affected / at risk) | 4/4 | 6/7 | 3/3 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cixutumumab Cohort 1 (N=4) | Cixutumumab Cohort 2 (N=7) | Cixutumumab Cohort 3 (N=3) | Cixutumumab Cohort 4 (N=7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Movement disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cixutumumab Cohort 1 (N=4) | Cixutumumab Cohort 2 (N=7) | Cixutumumab Cohort 3 (N=3) | Cixutumumab Cohort 4 (N=7)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (5) | 0 (0) | 1 (1)
Injection site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Blood amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 4 (8) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 2 (2) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days